CLINICAL TRIAL: NCT01682187
Title: Phase 1 Dose-Escalation Study of LY2157299 Monotherapy and in Combination With Lomustine in Patients With Recurrent Malignant Glioma
Brief Title: A Dose-Escalation Study in Participants With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8660; H9H-MC-JBAH (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — LY-2157299; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2157299 (Part A) (Experimental): Administered orally by tablet twice daily for two weeks followed by two weeks of no treatment for two 28-day cycles. Part A dose escalation will have starting dose of 40 mg/day and may increase up to 360 mg/day.
  Interventions: Drug: LY2157299
- LY2157299 + Lomustine (Part B) (Experimental): LY21547299 will be administered orally by tablet twice daily for two weeks followed by two weeks of no treatment for two 28-day cycles. Part B dose expansion will have starting dose of 80 mg twice daily and may increase up to 150 mg twice daily.
  Lomustine will be administered orally by capsule once on Day 7 of Cycle 1 after receiving LY2157299, and once after receiving LY2157299 on Day 21 of Cycles 2, 5, 8, 11, and every 4th cycle thereafter.
  Interventions: Drug: LY2157299; Drug: Lomustine

INTERVENTIONS:
Drug: LY2157299 — Administered orally
Drug: Lomustine — Administered orally
  Arms: LY2157299 + Lomustine (Part B)

SUMMARY:
This is a study of oral LY2157299 as monotherapy and in combination with lomustine in participants with recurrent malignant glioma.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Have histological or cytological evidence of relapsed malignant glioma (such as glioblastoma multiforme, anaplastic astrocytoma, anaplastic oligodendroglioma) for which no treatment of higher priority exists

  * Available baseline tumor specimen is required prior to considering participant to be enrolled. The original diagnostic tumor tissue is sufficient for this inclusion criteria, but where possible, freshly obtained tumor biopsy material may be obtained
  * Measurable disease to allow assessment of tumor response based on radiographic assessment following Macdonald criteria and Response Evaluation Criteria In Solid Tumors (RECIST)
* Have sufficient hepatic, renal, and hematological function
* Have a performance status of ≤2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy or other investigational therapy for at least 30 days prior to study enrollment and recovered from the acute effects of therapy
* Able to swallow tablets and capsules
* For females, reproductive potential must be either terminated (by surgery, radiation, or menopause) or attenuated by the use of an approved contraceptive method (including intrauterine or barrier devices) during and for 3 to 6 months after the study
* Male participants must be willing to use contraception during and for 3 to 6 months after the study

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Have moderate or severe cardiac disease:

  * Have the presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension
  * Have documented major electrocardiogram (ECG) abnormalities at the investigator's discretion (for example, symptomatic or sustained atrial or ventricular arrhythmias, second- or third-degree atrioventricular block, bundle branch blocks, ventricular hypertrophy, or recent myocardial infarction)
  * Have major abnormalities documented by echocardiography with Doppler (for example, moderate or severe heart valve function defect and/or left ventricular ejection fraction (LVEF) <50%, evaluation based on the institutional lower limit of normal)
  * Have predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress (for example, family history of aneurysms, Marfan syndrome, bicuspid aortic valve, evidence of damage to the large vessels of the heart documented by computerized tomography [CT] scan with contrast)
* Have current acute or chronic leukemia
* Women who are pregnant or lactating
* Have received prior nitrosourea (including lomustine) therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-12-15 (Actual); Primary Completion 2012-05-22 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Recommended Dose for Phase 2 Studies | Time of first dose to time of last dose (estimated up to 8 years)

SECONDARY OUTCOMES:
Number of Participants with Tumor Response | Time of first dose to time of last dose (estimated up to 8 years)
Biologically Effective Dose Range | Baseline, Days 1, 12, 13 of Cycle 1, Days 1 and 12 of Cycle 2 of Part A - LY2157299 as monotherapy
Pharmacokinetics (PK): Area Under the Concentration-Time Curve (AUC) | Part A Cycle 1: predose, up to 6 hours on Days 1, 3, 6, 12, 13, and 14; Part A Cycle 2: predose up to 6 hours on Days 1, 12, and 13. Part B Cycle 1: predose up to 6 hours on Days 1, 6, 7, 10, 12, 13, and 14
Pharmacokinetics (PK): Maximum Concentration (Cmax) | Part A Cycle 1: predose, up to 6 hours on Days 1, 3, 6, 12, 13, and 14; Part A Cycle 2: predose up to 6 hours on Days 1, 12, and 13. Part B Cycle 1: predose up to 6 hours on Days 1, 6, 7, 10, 12, 13, and 14

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland, United States
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville